CLINICAL TRIAL: NCT00652041
Title: Thalidomide-Cyclophosphamide-Dexamethasone in Patients < 75 Years or Velcade-Melfalan-Prednisone (V-MP)/Thalidomide-Cyclophosphamide-Dexamethasone in Patients >75 Years, in Refractary or Relapsed Multiple Myeloma
Brief Title: Bortezomib/Adriamycine/Melfalan/Prednisone (VAMP)/Thalidomide/Cyclophosphamide/Dexamethasone (TaCyDex) or Bortezomib/Melfalan/Prednisone (V-MP)/TaCyDex) in Refractary or Relapsed Multiple Myeloma
Acronym: TaCyDexVMP7
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, Pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TaCyDexVMP7
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed; Refractary
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Induction: 6 alternating cycles Bortezomib-Melfalan-Prednisone or Bortezomib- Adriamycine-Melfalan-Prednisone and Thalidomide-Cyclophosphamide-Dexamethasone, followed by other 6 maintenance cycles
  Interventions: Drug: Bortezomib; Drug: Thalidomide

INTERVENTIONS:
Drug: Bortezomib — Bortezomib, 1,3 mg/ m2 iv twice a week in combination with Melfalán 9 mg/m2 oral, days 1 to 4 and Prednisone, 60 mg/m2 oral, days 1 to 4
Drug: Thalidomide — Thalidomide, day 1 cycle 1, 100 mg/24 h. oral, in combination with cyclophosphamide and dexamethasone. If toxicity is <Grade 2, dose should be increased to 200 mg/24 h. in day 15
Drug: Bortezomib — Bortezomib, 1,3 mg/ m2 iv twice a week in combination with Melfalán 9 mg/m2 oral, days 1 to 4, Prednisone, 60 mg/m2 oral, days 1 to 4 and Adriamicine, 40 mg/m2 IV day 1 or Caelyx 30 mg/m2 IV day 1.

SUMMARY:
Multicentric study, open, single arm, designed to evaluate the efficacy(response rate and response duration) and security of a sequential scheme of treatment with Bortezomib in combination with Melfalan and Prednisone (V-MP) (patients > 75 years) or Bortezomib and Adriamycine in combination with Melfalan and Prednisone (VAMP) (patients <= 75 years) follow by Thalidomide in combination with Cyclophosphamide and Dexamethasone (TaCyDex) in patients with refractary or relapse multiple myeloma.

DETAILED DESCRIPTION:
Multicentric study, open, single arm, designed to evaluate the efficacy(response rate and response duration) and security of a sequential scheme of treatment with Bortezomib in combination with Melfalan and Prednisone (V-MP) (patients > 75 years) or Bortezomib and Adriamycine in combination with Melfalan and Prednisone (VAMP) (patients <= 75 years) follow by Thalidomide in combination with Cyclophosphamide and Dexamethasone (TaCyDex) in patients with refractary or relapse multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractary or relapsed multiple myeloma
* ECOG ≤ 3
* Life expectancy > 3 months
* Neutrophils account ≥ 0.5 X 10^9/L, platelets ≥ 30 X 10^9/L.
* Transaminases <3 times upper normal limit, bilirubin < 2 times upper normal limit
* Age > 18 years
* Time after last chemotherapy or radiotherapy > 1 month or time after transplantation > 2 months.
* No possible other actual treatment
* Written consent form

Exclusion Criteria:

* Candidate to second transplantation
* No following criteria
* Other neoplasties
* Peripheral neuropathy > Grade 2.
* Previous ileus paralytic
* Hepatic failure
* No controlled infection
* No controlled high calcium levels
* Any organic insufficiency that no permit follow the correct treatment
* Pregnancy, breast feeding or fertility without anticonceptive method
* Any psychological, social and/or familiar event that no permit follow the correct treatment
* Diabetes mellitus not controled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of a sequential scheme treatment with Bortezomib, Melfalan,Prednisone (V-MP) or Bortezomib, Adriamycine, Melfalan,Prednisone (VAMP) followed by Thalidomide, Cyclophosphamide and Dexamethasone (TaCyDex) in relapsed or refractory MM patients | 1 year

SECONDARY OUTCOMES:
Evaluate the response type in function to different initial situation (primary resistance, relapse, progression) | 1 year
To analyze the response duration | 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Morales Messeguer, Murcia
  - Hospital Virgen de la Vega, Murcia
  - Hospital de la Diputación de Navarra, Navarra
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital La Fe, Valencia

REFERENCES:
- See also: spanish hematology association — http://aehh.org